CLINICAL TRIAL: NCT04504383
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled, Parallel-group, Multi-center Study to Evaluate the Safety and Efficacy of Oral PN-943 in Subjects With Moderate to Severe Active Ulcerative Colitis
Brief Title: PN-943 in Adults With Moderate to Severe Active Ulcerative Colitis (UC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Protagonist Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PN-943-03
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Ulcerative Colitis Chronic Moderate; Ulcerative Colitis Chronic Severe
Keywords: Inflammatory Bowel Disease (IBD)
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: 12-week randomized, double-blind, placebo-controlled, parallel design study in patients with moderate to severe active UC. It will be followed by 40 weeks of Extended Active Treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PN-943 450 mg BID (Experimental): Oral administration of PN-943 450 mg BID
  Interventions: Drug: PN-943
- PN-943 150 mg BID (Experimental): Oral administration of PN-943 150 mg BID
  Interventions: Drug: PN-943
- Placebo BID (Placebo Comparator): Oral administration of matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PN-943 — Administered by the oral route BID for the duration of the study.
  Arms: PN-943 150 mg BID; PN-943 450 mg BID
Drug: Placebo — Administered by the oral route BID for 12 weeks.
  Arms: Placebo BID

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and clinical efficacy of PN-943 450 mg twice daily [BID] and PN-943 150 mg BID, compared with placebo BID, in subjects with moderate to severe active Ulcerative Colitis (UC).

DETAILED DESCRIPTION:
The study consists of a 12-week double-blind, placebo-controlled treatment period. Participants will be randomized in a 1:1:1 ratio to PN-943 450 mg BID, PN-943 150 mg BID, or matching placebo BID.

Participants who successfully complete the double-blind period may be eligible for an extended treatment period of 40 weeks duration.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and female subjects age 18 (or the minimum country specific age of consent if >18) to 75 years.
2. Subject understands the study procedures and agrees to participate in the study by giving written informed consent.
3. Diagnosis of UC supported by appropriate documentation of biopsy results consistent with UC.
4. Moderate to severe active UC.
5. Demonstrated inadequate response, loss of response, or intolerance of at least 1 of oral aminosalicylates (5-ASAs), corticosteroids, immunomodulators, or a biologic (excluding vedolizumab).

Key Exclusion Criteria:

1. Subject with a current diagnosis of Crohn's disease (CD), indeterminate colitis (IC), microscopic colitis, ischemic colitis, radiation colitis.
2. History of colonic dysplasia other than completely removed low-grade dysplastic lesion.
3. History of active bacterial, viral, fungal or mycobacterial infection requiring hospitalization or IV antibiotic/anti-infective treatment within 4 weeks of screening or oral antibiotics/anti-infectives within 2 weeks of screening.
4. Prior treatment with vedolizumab, natalizumab, or any agent targeting the α4β7 or β1 integrin or planned during the study.
5. Positive stool test for C. difficile.
6. Chronic recurrent or serious infection.
7. Known primary or secondary immunodeficiency.
8. Pregnant or lactating female or considering becoming pregnant during the study or within 30 days after the last dose of study medication.
9. History of any major neurological disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving clinical remission at Week 12 compared to placebo. | Week 12
  Clinical remission is determined using the Adapted Mayo score (sum of 3 subscores from the Mayo score):
  * Stool frequency subscore (SFS)
  * Rectal bleeding subscore (RBS)
  * Endoscopic subscore (ESS)

SECONDARY OUTCOMES:
Comparison between PN-943 high-dose and low-dose individually to placebo. | Week 12
  1. Proportion of subjects with endoscopic improvement.
  2. Proportion of subjects achieving endoscopic remission.
  3. Proportion of subjects with histological improvement.
  4. Proportion of subjects achieving histological remission.
  5. Proportion of subjects with mucosal healing.

OTHER OUTCOMES:
Proportion of subjects achieving clinical remission at Week 52. | Week 52
  Clinical remission is determined using the Adapted Mayo score (sum of 3 subscores from the Mayo score):
  * Stool frequency subscore (SFS)
  * Rectal bleeding subscore (RBS)
  * Endoscopic subscore (ESS)

CONTACTS AND LOCATIONS:
Locations (94):
- United States (29):
  - Protagonist Investigational Site, Tucson, Arizona
  - Protagonist Investigational Site, Garden Grove, California
  - Protagonist Investigational Site, Los Angeles, California
  - Protagonist Investigational Site, Murrieta, California
  - Protagonist Investigational Site, San Francisco, California
  - Protagonist Investigational Site, Colorado Springs, Colorado
  - Protagonist Investigational Site, Kissimmee, Florida
  - Protagonist Investigational Site, Miami, Florida
  - Protagonist Investigational site, Orlando, Florida
  - Protagonist Investigational Site, Saint Augustine, Florida
  - Protagonist Investigational Site, Wesley Chapel, Florida
  - Protagonist Investigational Site, Metairie, Louisiana
  - Protagonist Investigational Site, Glen Burnie, Maryland
  - Protagonist Investigational Site, Chesterfield, Michigan
  - Protagonist Investigational Site, Troy, Michigan
  - Protagonist Investigational Site, Jackson, Mississippi
  - Protagonist Investigational Site, St Louis, Missouri
  - Protagonist Investigational Site, Englewood, New Jersey
  - Protagonist Investigational Site, North Massapequa, New York
  - Protagonist Investigational Site, Charlotte, North Carolina
  - Protagonist Investigational Site, Norman, Oklahoma
  - Protagonist Investigational Site, Oklahoma City, Oklahoma
  - Protagonist Investigational Site, Orangeburg, South Carolina
  - Protagonist Investigational Site, Nashville, Tennessee
  - Protagonist Investigational Site, Austin, Texas
  - Protagonist Investigational site, Garland, Texas
  - Protagonist Investigational Site, Pasadena, Texas
  - Protagonist Investigational Site, Spring, Texas
  - Protagonist Investigational site, Lynchburg, Virginia
- Austria (3):
  - Protagonist Investigational Site, Innsbruck
  - Protagonist Investigational Site, Salzburg
  - Protagonist Investigational Site, Vienna
- Protagonist Investigational Site, Sofia, Bulgaria
- Canada (6):
  - Protagonist Investigational Site, Kelowna, British Columbia
  - Protagonist Investigational Site, Vancouver, British Columbia
  - Protagonist Investigational Site, West Vancouver, British Columbia
  - Protagonist Investigational Site, North Bay, Ontario
  - Protagonist Investigational Site, Toronto, Ontario
  - Protagonist Investigational Site, Vaughan, Ontario
- Protagonist Investigational Site, Tbilisi, Georgia
- Germany (3):
  - Protagonist Investigational Site, Berlin
  - Protagonist Investigational Site, Kiel
  - Protagonist Investigational Site, Tübingen
- Hungary (3):
  - Protagonist Investigational Site, Budapest
  - Protagonist Investigational Site, Debrecen
  - Protagonist Investigational Site, Székesfehérvár
- Italy (6):
  - Protagonist Investigational Site, Castellana Grotte
  - Protagonist Investigational Site, Modena
  - Protagonist Investigational Site, Negrar
  - Protagonist Investigational Site, Padua
  - Protagonist Investigational Site, Roma
  - Protagonist Investigational Site, San Giovanni Rotondo
- Poland (19):
  - Protagonist Investigational Site, Poznan, Greater Poland Voivodeship
  - Protagonist Investigational Site, Bydgoszcz
  - Protagonist Investigational Site, Częstochowa
  - Protagonist Investigational Site, Katowice
  - Protagonist Investigational Site, Krakow
  - Protagonist Investigational Site, Ksawerów
  - Protagonist Investigational Site, Lodz
  - Protagonist Investigational Site, Lublin
  - Protagonist Investigational Site, Nowy Targ
  - Protagonist Investigational Site, Piotrkow Trybunalski
  - Protagonist Investigational Site, Poznan
  - Protagonist Investigational Site, Rzeszów
  - Protagonist Investigational Site, Sopot
  - Protagonist Investigational Site, Swidnica
  - Protagonist Investigational Site, Torun
  - Protagonist Investigational Site, Tychy
  - Protagonist Investigational Site, Warsaw
  - Protagonist Investigational Site, Wroclaw
  - Protagonist Investigational Site, Włocławek
- Russia (11):
  - Protagonist Investigational Site, Chelyabinsk
  - Protagonist Investigational Site, Moscow
  - Protagonist Investigational Site, Novosibirsk
  - Protagonist Investigational Site, Perm
  - Protagonist Investigational Site, Pyatigorsk
  - Protagonist Investigational Site, Saint Petersburg
  - Protagonist Investigational Site, Samara
  - Protagonist Investigational Site, Saratov
  - Protagonist Investigational Site, Stavropol
  - Protagonist Investigational Site, Tomsk
  - Protagonist Investigational Site, Tyumen
- Protagonist Investigational Site, Zrenjanin, Serbia
- South Korea (5):
  - Protagonist Investigational Site, Busan
  - Protagonist Investigational Site, Daegu
  - Protagonist Investigational Site, Daejeon
  - Protagonist Investigational Site, Seoul
  - Protagonist Investigational site, Seoul
- Ukraine (6):
  - Protagonist Investigational Site, Ivano-Frankivsk
  - Protagonist Investigational Site, Kherson
  - Protagonist Investigational Site, Kyiv
  - Protagonist Investigational Site, Lviv
  - Protagonist Investigational Site, Vinnytsia
  - Protagonist Investigational Site, Zhytomyr

IPD SHARING:
Plan to Share IPD: No